CLINICAL TRIAL: NCT03193723
Title: Efficacy of Ultrasound Guided Local Anesthetic Field Block (A Five Step Procedure) as a Sole Anesthetic for Open Inguinal Hernia Repair Versus Spinal Anesthesia: A Randomized Controlled Study.
Brief Title: Ultrasound Guided Local Anesthetic Field Block (A Five Step Procedure) for Open Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eslam Ayman Mohamed Shawki (Other)
Responsible Party: Sponsor-Investigator, Eslam Ayman Mohamed Shawki, Lecturer of anesthesia, SICU & Pain Management, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UsHernia
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Inguinal Hernia
Keywords: Hernia; Local anesthesia; ultrasound
MeSH Terms: conditions — Hernia, Inguinal; Hernia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): US guided five step field block will be performed
  Interventions: Procedure: US guided five step field block
- Group B (Active Comparator): Spinal anesthesia will be administered in sitting position
  Interventions: Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: US guided five step field block — Ultrasound will guide needle insertion in the following layers (except intradermic injection):
  * Subdermic infiltration. Approximately 8 milliliters
  * Intradermic injection (making of the skin wheal). of approximately 6 milliliters.
  * Deep subcutaneous injection. 8 milliliters of the mixture will be injected deep into the subcutaneous adipose
  * Subfascial infiltration. Approximately eight milliliters of the anesthetic mixture will be injected immediately underneath the aponeurosis of the external oblique.
  * Pubic tubercle and hernia sac injection. Occasionally, infiltration of ten milliliters of the mixture at the level of the pubic tubercle, around the neck and inside the indirect hernia sac
  Arms: Group A
Procedure: Spinal anesthesia — Spinal anesthesia will be administered in sitting position, with 25 gauge Quincke spinal needle in L3-L4 intervertebral space, under all aseptic precautions and local infiltration, with 3.0 ml of 0.5% bupivacaine (heavy) after ensuring free, clear and adequate flow of cerebrospinal fluid. After giving spinal anesthesia, patient will be made to lie supine.
  Arms: Group B

SUMMARY:
The aim of this study is to evaluate success, efficacy, feasibility and safety of a simple five step ultrasound guided local anesthetic infiltration technique for unilateral open inguinal hernia repair and to determine the non-inferiority of the block to spinal anesthesia by comparing intraoperative and postoperative complications, pain control and patient and surgeon satisfaction of the block with spinal anesthesia.

DETAILED DESCRIPTION:
Open Inguinal hernia repair is one of the commonest procedures performed worldwide. Still, there is no consensus regarding the optimum anesthesia technique for this surgery. General, spinal, epidural and local anesthesia techniques have all been used, each having its own advantages and disadvantages.

General anesthesia carries risks of possible airway complications, postoperative deterioration of cognitive function, sore throat, nausea, vomiting and prolonged period of immobilization with associated risk of deep vein thrombosis and longer hospital stay. Spinal anesthesia, although effective, is not without risk in patients with decompensated heart disease, recent head injury, convulsions and coagulopathies. Also spinal and epidural anesthesia have been associated with hemodynamic instability, vomiting, urinary retention, post-dural puncture headache, and backache.

Use of pre-incision infiltration of local anesthetics for field blocks has been found to be an effective adjunct as well as an alternative to spinal and general anesthesia in many studies. Combined with sedation or on its own, it offers less cardiovascular instability, early ambulation and effective post-operative pain control. Also, it has been found to reduce hospital costs by 50% and gives better patient satisfaction.

Harvey Cushing and William Halsted first described the inguinal field block in 1900. since then, its efficacy and advantages have been compared by many surgeons and anesthesiologists in a number of studies. Refinements and modifications in the technique still continue. In 1963, Joseph L Ponka described in great detail a seven step procedure of performing it in 837 patients successfully.

In 1994, Parvis and colleagues did a step by step technique for local anesthetic infiltration field block for open inguinal hernia repair.

Ultrasonography is a safe and effective form of imaging. Over the past two decades, ultrasound equipment has become more compact, of higher quality and less expensive. Ultrasounds have been used to guide needle insertion and a number of approaches to nerves and plexuses have been reported. A clear advantage of the technique is that ultrasound produces "living pictures" or "real-time" images. The identification of neuronal and adjacent anatomical structures (blood vessels, peritoneum, bone, organs) along with the needle is another advantage. Moreover, anatomical variability may be responsible for block failures, and ultrasound technology enabling direct visualization may overcome this problem. Sonographic visualization allows for the performance of extra-epineurial needle tip positioning and administration of local anesthetic avoiding intra-epineurial injection.

A modification to the technique performed by Parvis and colleagues will be tested in this study. Our modification will be performing the technique under ultrasound guidance and completely before skin incision, which, to the best of our knowledge, was not attempted in the literature before.

Local anesthesia administered before skin incision produces longer postoperative analgesia because local infiltration theoretically inhibits the build-up of local nociceptive molecules and, therefore, there is better pain control in the postoperative period.This study aims at evaluating success, efficacy, feasibility and safety of a simple five step ultrasound guided local anesthetic infiltration technique for unilateral open inguinal hernia repair and also to compare intraoperative and postoperative complications and pain control of the block with spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA score I, II or Ш.
* Patients with unilateral inguinal hernia for elective open mesh repair hernioplasty operation.

Exclusion Criteria:

* Bilateral, recurrent or complicated inguinal hernia.
* Emergency operations or operation that lasts more than two hours.
* Patients with drug or alcohol abuse history.
* Chronic pain, with daily use of analgesics.
* Contraindication to local anesthesia.
* Contraindication of spinal anesthesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
NRS 4 hours postoperative | 4 hours
  Numerical Rating pain score 4 hours postoperative

SECONDARY OUTCOMES:
NRS 30 minutes postoperative | 30 minutes
  Numerical Rating pain score 30 minutes postoperative.
NRS 12 hours postoperative | 12 hours
  Numerical Rating pain score 12 hours postoperative.
Time of first rescue analgesic dose | 12 hours
  The time of request for the first rescue dose of analgesic medication
Total analgesic dose in the first 12 hours postoperative | 12 hours
  The total doses of analgesics needed (whether opioids or non-opioids) to maintain an NRS score < 3 over the first 12 hours post-operative
Incidence of Side effects | 12 hours
  Complications including nausea, vomiting, wound hematoma, hypotension, persistent headache and urinary retention
Time for ambulation | 12 hours
  The time needed to start pain free unassisted ambulation and the duration of hospital stay.
Intra operative patient satisfaction | 12 hours
  Intra operative patient satisfaction (rated as 1 to be very satisfied, 2 moderately satisfied and 3 poorly satisfied.)
Intra operative surgeon satisfaction | 12 hours
  Intra operative surgeon satisfaction with the type of anesthesia (satisfied or not)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo University teaching hospitals (Kasr Alainy), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anand A, Sinha PA, Kittappa K, Mulchandani MH, Debrah S, Brookstein R. Review of Inguinal Hernia Repairs by Various Surgical Techniques in a District General Hospital in the UK. Indian J Surg. 2011 Jan;73(1):13-8. doi: 10.1007/s12262-010-0156-7. Epub 2011 Jan 8. PMID 22211031
- [Background] Santos Gde C, Braga GM, Queiroz FL, Navarro TP, Gomez RS. Assessment of postoperative pain and hospital discharge after inguinal and iliohypogastric nerve block for inguinal hernia repair under spinal anesthesia: a prospective study. Rev Assoc Med Bras (1992). 2011 Sep-Oct;57(5):545-9. doi: 10.1590/s0104-42302011000500013. English, Portuguese. PMID 22012289
- [Background] Flanagan L Jr, Bascom JU. Repair of the groin hernia. Outpatient approach with local anesthesia. Surg Clin North Am. 1984 Apr;64(2):257-67. doi: 10.1016/s0039-6109(16)43283-4. PMID 6729669
- [Background] Belavy D, Cowlishaw PJ, Howes M, Phillips F. Ultrasound-guided transversus abdominis plane block for analgesia after Caesarean delivery. Br J Anaesth. 2009 Nov;103(5):726-30. doi: 10.1093/bja/aep235. Epub 2009 Aug 22. PMID 19700776
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Chanthong P, Abrishami A, Wong J, Herrera F, Chung F. Systematic review of questionnaires measuring patient satisfaction in ambulatory anesthesia. Anesthesiology. 2009 May;110(5):1061-7. doi: 10.1097/ALN.0b013e31819db079. PMID 19352161
- [Background] Prakash D, Heskin L, Doherty S, Galvin R. Local anaesthesia versus spinal anaesthesia in inguinal hernia repair: A systematic review and meta-analysis. Surgeon. 2017 Feb;15(1):47-57. doi: 10.1016/j.surge.2016.01.001. Epub 2016 Feb 16. PMID 26895656